CLINICAL TRIAL: NCT01916616
Title: A Multidisciplinary Approach to Vocal Cord Dysfunction: A Novel Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CAMC Health System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1997292
Record Dates: First submitted 2013-08-01; First posted 2013-08-05 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Vocal Cord Dysfunction
Keywords: paradoxical vocal fold motion; cognitive-behavioral therapy
MeSH Terms: conditions — Vocal Cord Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Four therapy sessions with a psychologist utilizing cognitive-behavioral therapy techniques — At the four therapy sessions, subjects will work with the psychologist to identify the triggers of their VCD episodes, learn to self-monitor symptoms and reactions, and be taught breathing retraining/relaxation techniques. The goal is to decrease patterns of subjects' thinking or behaviors that exacerbate distress from VCD symptoms.

SUMMARY:
Vocal Cord Dysfunction (VCD) is characterized by involuntary closure of the vocal cords while inhaling. Children and adolescents with VCD may experience multiple symptoms, including difficulty breathing, coughing, wheezing, neck tightness, and voice changes. There is limited information on optimal management of VCD. In our proposed study, we will use cognitive-behavioral therapy (CBT) techniques to change how patients respond to their VCD symptoms. Measurements of airflow during breathing as well as symptom frequency and intensity will be examined prior to and following a series of four therapy sessions with a clinical psychologist that are focused on teaching patients strategies to decrease symptom reactivity.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent patients presenting to West Virginia University, Charleston Division Sub-specialty Clinic for Pediatric Pulmonology with a clinical diagnosis of vocal cord dysfunction.
* Diagnosed with VCD within 12 months prior to study enrollment. between the ages of 13 and 18 years old.
* Currently symptomatic for VCD.
* Must have a baseline PFT to reference at the time of diagnosis. Additionally in patients who were diagnosed with VCD 6 months or more prior to study enrollment, current PFT results as part of routine care, are required.
* A parent or guardian must agree to participate in the four behavioral therapy sessions with his or her child.

Exclusion Criteria:

* Severe psychiatric disorders (ex. psychosis, suicidal ideation)
* Developmental delay
* Previous speech therapy for the treatment of VCD.
* Currently receiving psychological counseling.
* In open Child Protective Services cases.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2013-09-01 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2015-06-30 (Actual)

PRIMARY OUTCOMES:
Change in frequency and intensity of VCD symptoms | Post intervention at 1 to 3 weeks
  Self-reported number of symptomatic episodes and mean intensity of episodes pre and post-CBT intervention will be compared. Symptom intensity will be measured using an 11 point Likert Scale for self-reported distress for each recorded VCD episode.

SECONDARY OUTCOMES:
Change in pulmonary function testing (PFT) measures | Post intervention at 1 to 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Maupin, MD, Principal Investigator — WVU Charleston Division
Locations (1):
- Department of Pediatric, West Virginia University-Charleston Division, Charleston, West Virginia, United States